CLINICAL TRIAL: NCT01892709
Title: Efficacy of an Acute Pain Titration Protocol Driven by Patient Response to a Simple Query: Do You Want More Pain Medication?
Brief Title: Titration of Intravenous Hydromorphone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-12-408
Record Dates: First submitted 2013-06-06; First posted 2013-07-04 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Acute Severe Pain
Keywords: acute; pain; emergency department; hydromorphone; in ER
MeSH Terms: conditions — Pain; Emergencies | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydromorphone (Experimental): All eligible patients will receive 1 mg IV hydromorphone. Thereafter, they will be repeatedly asked the question, "Do you want more pain medicine?" This question will be asked 30 minutes after they answered "no" or 30 minutes after the completion of the next dose of 1 mg IV hydromorphone, which occurs when the patients answers "yes". Patients will receive a maximum of 4 mg IV hydromorphone over a 4 hour period.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone
  Other Names: Dilaudid

SUMMARY:
This is an exploratory, hypothesis-generating safety and efficacy study for patients who come to the ER in acute (less than 7 days in duration) severe pain. Patients with chronic pain will not be enrolled. Eligible patients will receive up to a maximum of 4 mg IV hydromorphone over a 4 hour period. Hydromorphone will be given as 1 mg increments based on how the patient responds to the question, "Do you want more pain medicine?". This question will be asked repeatedly 30 minutes after the patient answers "no" or 30 minutes after the most recent dose of IV hydromorphone (which occurs if the patient answers "yes"). Up to 10% (approximately 30 patients) will serve as a pilot at the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age greater than 21 years: Patients under the age of 21 are automatically triaged to the Children's Hospital at Montefiore Emergency Department, and hence cannot be enrolled in this study.

  2. Age less than 65 years: Patients age 65 and over will be excluded from this study as the effects on opioids on the elderly may be different than in the non-elderly.

  3. Pain with onset within 7 days: Pain within seven days is the definition of acute pain that has been used in Emergency Department (ED) literature.

  4. ED attending physician's judgment that patient's pain warrants use of morphine

  5. Normal mental status: In order to provide measures of pain experienced the patient needs to have a normal mental status. Orientation to person, place and time will be used as an indicator of sufficiently normal mental status to participate in the study.

Exclusion Criteria:

* 1. Prior use of methadone: the effect of methadone use on the perception of acute pain is unknown and suspected to be altered. Similar to sickle cell patients and chronic cancer patients, patients on methadone usually require significantly higher doses of opioids to control their pain.

  2. Use of other opioids or tramadol within past 24 hours: to avoid introducing bias related to opioid tolerance that may alter the response to the study medication thereby masking the medication's effect.

  3. Prior adverse reaction to hydromorphone: patients will be excluded if they state that they have an allergy to hydromorphone.

  4. Chronic pain syndrome: frequently recurrent or daily pain for at least 3 months result in alteration in pain perception which is thought to be due to down-regulation of pain receptors. Examples of chronic pain syndromes include sickle cell anemia, osteoarthritis, fibromyalgia, migraine, and peripheral neuropathies.

  5. Patients for whom the attending physician suspects is addicted to opioids: patients will be excluded if the attending suspects the patient may be addicted to opioids or seeking to obtain them for diversionary reasons, such as for monetary profit or other illicit use.

  6. Alcohol intoxication: the presence of alcohol intoxication as judged by the treating physician may alter perception, report, and treatment of pain.

  7. Systolic Blood Pressure <100 mm Hg: Hydromorphone can produce peripheral vasodilation that may result in orthostatic hypotension or syncope.

  8. Respiratory rate < 12/minute: Hydromorphone can cause respiratory depression.

  9. Oxygen saturation <95% on room air: For this study, oxygen saturation must be 95% or above on room air in order to be enrolled.

  10. Heart rate < 60 beats/minute: Hydromorphone can cause bradycardia.

  11. Use of monoamine oxidase (MAO) inhibitors in past 30 days: MAOs have been reported to intensify the effects of at least one opioid drug causing anxiety, confusion and significant respiratory depression or coma.

  12. Carbon dioxide measurement greater than 46: three subsets of patients will have their carbon dioxide measured using a handheld capnometer prior to enrollment in the study. If the carbon dioxide measurement is greater than 46, then the patient will be excluded from the study. The 3 subsets are as follows:
  1. All patients who have a history of chronic obstructive pulmonary disease (COPD)
  2. All patients who report a history of asthma together with greater than a 20 pack-year smoking history
  3. All patients reporting less than a 20 pack-year smoking history who are having an asthma exacerbation

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew K Chang, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center Moses Emegency Department, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydromorphone: All eligible patients will receive 1 mg IV hydromorphone. Thereafter, they will be repeatedly asked the question, "Do you want more pain medicine?" This question will be asked 30 minutes after they answered "no" or 30 minutes after the completion of the next dose of 1 mg IV hydromorphone, which occurs when the patients answers "yes". Patients will receive a maximum of 4 mg IV hydromorphone over a 4 hour period.
  Hydromorphone
Period: Overall Study
Arm/Group | Hydromorphone
Started | 215
Completed | 215
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 8 patients excluded from initial 215 for protocol violations: 1 from missing data, 7 for failure to receive intravenous hydromorphone after requesting it
Arm/Group | Hydromorphone
Number analyzed (Participants) | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 143
  Black | 44
  White/Other | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 207
Weight [Mean (Standard Deviation); unit: lbs] | 177 (34)
Location of pain [Count of Participants; unit: Participants]
  Abdomen/pelvis | 153
  Flank | 22
  Back | 15
  Extremities | 8
  Other | 9
Initial NRS pain intensity [Count of Participants; unit: Participants] — Pain intensity is measured on the numerical rating scale (NRS) from 0 ("no pain") to 10 ("worst pain imaginable")
  Participants
    NRS = 5-7 | 21
    NRS = 8 | 27
    NRS = 9 | 41
    NRS = 10 | 118
Nauseated or vomited before receiving first dose of opioid [Count of Participants; unit: Participants] | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requesting Pain Medication in Different Patterns Over Time
Description: This is a descriptive hypothesis-generating trial, which is why it is not being compared in a randomized fashion to a comparison group. We are examining extended titration by expanding our "1+1" protocol to a "1+1+1+1" protocol and the various patterns of opioid request. For example, some may state "no" every time they are asked "Do you want more pain medication?" Some will state "yes" each time, and others will answer "yes" and "no" at different time periods. We will report these various patterns (i.e. X participants answered "no" everytime they were asked, Y answered "yes" everytime they were asked, Z answered "no" twice, etc).
  Time points 2, 3, and 4 are dependent on patient response to "Do you want more pain medication?" Time 1 is 30 min post-baseline. For those who answer "no", Time 2 is 30 minutes later (at 1 hour), and for yes, Time 2 is 30 minutes after additional pain medication is given. This pattern follows for Time 3 and 4, with a total study time of 4 hours
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 207
Participants
  No requests for additional pain medication | 94
  Requested additional pain medication, Time 1 only | 20
  Requested additional pain medication, Time 2 only | 22
  Requested additional pain medication, Time 3 only | 19
  Requested additional pain medication, Time 4 only | 18
  Requested add'l pain medication at >1 time point | 2

2. Secondary Outcome: Adverse Events and Side Effects by Total Amount of Hydromorphone Received
Time Frame: 120 min
Population: Nausea and vomiting were only assessed as adverse events among patients who did not have nausea and vomiting before the study began
Measure: Count of Participants; unit: Participants
Groups:
- 1 mg Hydromorphone: Received 1 mg of IV hydromorphone, and answered "no" to all repeated questions of "Do you want more pain medication?"
- 2 mg Hydromorphone: Received 2 mg of IV hydromorphone, in 2 1-mg doses.
- 3 mg Hydromorphone: Received 3 mg of IV hydromorphone, in 3 1-mg doses
- 4 mg Hydromorphone: Received 4 mg of IV hydromorphone, in 4 1-mg doses
Arm/Group | 1 mg Hydromorphone | 2 mg Hydromorphone | 3 mg Hydromorphone | 4 mg Hydromorphone
Number analyzed (Participants) | 114 | 78 | 9 | 6
Participants
  Oxygen saturation <95% | 3 | 5 | 1 | 0
  Respiratory Rate <10 breaths/min | 1 | 0 | 1 | 0
  Pulse rate <50 beats/min | 1 | 1 | 0 | 0
  Systolic blood pressure <90 mmHg | 1 | 0 | 0 | 0
  Pruritus | 8 | 8 | 2 | 2
  Nausea: number analyzed (Participants) | 28 | 26 | 2 | 4
  Nausea | 6 | 14 | 2 | 3
  Vomiting: number analyzed (Participants) | 28 | 26 | 2 | 4
  Vomiting | 4 | 5 | 0 | 0

3. Post Hoc Outcome: Number of Patients Responding to the Question, "Do You Want More Pain Medication?" at Each Time Point
Description: Time points 2, 3, and 4 are dependent on patient response to "Do you want more pain medication?" Time 1 is 30 min post-baseline. For those who answer "no" at Time 1, Time 2 is 30 minutes later (at 1 hour), and for those who answer yes, Time 2 is 30 minutes after additional pain medication is given. This pattern follows for Time 3 and 4, with a total study time of 4 hours
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 207
Participants
  Time 1: Yes | 42
  Time 1: No | 165
  Time 2: Yes | 41
  Time 2: No | 166
  Time 3: Yes | 31
  Time 3: No | 176
  Time 4: Yes | 39
  Time 4: No | 168

4. Post Hoc Outcome: Mean Pain Intensity Score in Numerical Rating Scale (NRS) Units at Each Time Point, Based on Response to the Question, "Do You Want More Pain Medication?"
Description: Pain intensity is measured on the numerical rating scale (NRS) with scores from 0 ("no pain") to 10 ("worst pain imaginable").
  Time points 2, 3, and 4 are dependent on patient response to "Do you want more pain medication?" Time 1 is 30 min post-baseline. For those who answer "no" at Time 1, Time 2 is 30 minutes later (at 1 hour), and for those who answer yes, Time 2 is 30 minutes after additional pain medication is given. This pattern follows for Time 3 and 4, with a total study time of 4 hours
Time Frame: 4 hours
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 207
units on a scale
  Time 1, Yes | 7.4 [3 to 10]
  Time 1, No | 3.8 [0 to 10]
  Time 2, Yes | 7.2 [4 to 10]
  Time 2, No | 2.9 [0 to 7]
  Time 3, Yes | 7.1 [3 to 10]
  Time 3, No | 3.1 [0 to 10]
  Time 4, Yes | 6.8 [0 to 10]
  Time 4, No | 2.4 [0 to 8]

ADVERSE EVENTS:
Time Frame: 120 minutes
Arm/Group | Hydromorphone
All-Cause Mortality (participants affected / at risk) | 0/207
Serious Adverse Events (participants affected / at risk) | 0/207
Other Adverse Events (participants affected / at risk) | 68/207
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Hydromorphone (N=207)
Oxygen saturation <95% (Respiratory, thoracic and mediastinal disorders) | 9
Respiratory rate < 10 breaths/min (Respiratory, thoracic and mediastinal disorders) | 2
Pulse rate < 50 beats/min (Vascular disorders) | 2
Systolic blood pressure < 90 mmHg (Vascular disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 20
Nausea (Gastrointestinal disorders) | 25/60 — excluding patients who had nausea or vomiting before the study began
Vomiting (Gastrointestinal disorders) | 9/60 — excluding patients who had nausea or vomiting before the study began

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes